CLINICAL TRIAL: NCT01808456
Title: Phase IV, Pilot, Randomized, Investigator-blinded, Study to Evaluate the Reactogenicity and Immunogenicity of Standard-dose Versus High-dose Inactivated Influenza Vaccine After Kidney, Heart and Lung Transplantation.
Brief Title: Standard-dose Versus High-dose Flu Vaccine in Solid Organ Transplant.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IFH20132015
Record Dates: First submitted 2013-03-04; First posted 2013-03-11 (Estimated); Results first posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Influenza, Human; Transplantation Infection
Keywords: kidney transplant; heart transplant; lung transplant; influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Dose Flu Vaccine (Experimental): influenza trivalent inactive vaccine high dose. IM (intramuscular) injection one time administration
  Interventions: Biological: influenza trivalent inactive vaccine high dose
- Flu Vaccine (Active Comparator): influenza trivalent inactive vaccine IM injection one time administration
  Interventions: Biological: influenza trivalent inactive vaccine

INTERVENTIONS:
Biological: influenza trivalent inactive vaccine — one time IM injection of standard influenza vaccine to measure immunogenicity, safety, and efficacy in organ transplant recipients
  Other Names: Fluzone(R); flu vaccine
  Arms: Flu Vaccine
Biological: influenza trivalent inactive vaccine high dose — one time IM injection of high dose influenza vaccine to measure immunogenicity, safety, and efficacy in organ transplant recipients
  Other Names: Fluzone High Dose (R)
  Arms: High Dose Flu Vaccine

SUMMARY:
Influenza infection in recipients of solid organ transplants recipients while on maintenance immunosuppressant therapy is associated with increased morbidity and mortality. Although influenza vaccination is recommended in these high-risk patients, safety and immunogenicity of commercially available different strengths of influenza vaccine have not been established.

The primary study objective is to determine the safety and immunogenicity of Fluzone and Fluzone High-Dose, with a secondary objective to determine the tolerability and efficacy of two different strengths of trivalent influenza vaccine (TIV, flu vaccine). Both vaccines are commercially available for use in the general population. Fluzone is approved for use in 6 months of age and older, and Fluzone High-Dose is approved for use in 65 years of age and older.

This is an exploratory, open-label, parallel group, observer blinded, prospective study. All recipients of kidney, lung, heart transplants who attend for post-transplant follow-up, at least 30-days after transplantation at Inova Fairfax Hospital Transplant Center will be eligible for enrollment.

Enrolled patients will be followed for three months (a total of 4 visits) following enrollment and randomization: day 0 (enrollment) and follow-up visits at weeks 1, 4, 8, and 12.

DETAILED DESCRIPTION:
A potential strategy to enhance immune responses to influenza vaccine in this patient population could be to use different strengths of TIV. One of the pathways that can improve the immunogenicity of inactivated vaccines is to increase the dose of influenza antigens contained in the vaccine. Studies have demonstrated that increasing the dose of the influenza virus hemagglutinin for each of the commonly encountered viral strains beyond the conventional dose of 15 microgram for each strain is associated with dose-dependent increase in serum antibody titers.

Influenza TIV is commercially available in two different strengths, Fluzone as well as Fluzone High-Dose, and it is valuable because of variable immunogenic potency of different strengths. Fluzone is approved for use in persons 6 months of age and older. High-dose Fluzone is approved for use in persons 65 years of age and older.

The purpose of this exploratory study is to assess the safety, tolerability, and immunogenicity of these two commercially available different strengths of TIV in solid organ transplant recipients (kidney, heart and lung) in the period after 30 days after transplant procedure. We will evaluate the safety, tolerability (reactogenicity) and immunogenicity of two different strengths of commercially available TIV in a single center, cluster randomization, investigator blinded, study by enrolling patients in the post-transplant clinic at Inova Fairfax Hospital from: August 1, 2013 - March 31, 2014; and August 1, 2014 to March 31, 2015.

Study protocol will remain active till December 31, 2016. All bio-specimens will be stored till December 31, 2016.

ELIGIBILITY:
Inclusion Criteria:

1. All adults age ≥18 years of age following solid organ transplants (kidney, heart and lung) of all races and gender unless as specified in the exclusion criteria.
2. At least 30 days after organ transplantation of kidney, heart, or lung.
3. In good health as determined by a) medical history, b) physical examinations, c) clinical judgment of the investigator team.
4. Informed consent will be obtained from all the subjects before enrollment into the study, after the nature of the study has been fully explained to the satisfaction of the participant.
5. Non-English speaking persons will be included ONLY if consent can be obtained with the help of the translator or interpreter.

Exclusion Criteria:

1. Less than 30 days after transplantation procedure.
2. Post operative complications of any type.
3. Transplant organ dysfunction and/or under evaluation for possible infection.
4. Recent acute transplant rejection and treatment for rejection for the past 30 days.
5. Receiving another investigational drug or biologic for transplant.
6. Previous history of allergic reaction to influenza vaccine, chicken egg or other unknown allergic reactions to flu vaccine or other vaccines.
7. Acute ongoing respiratory illness.
8. Bleeding diathesis or on anticoagulation therapy.
9. Major surgery (pre-arranged) planned during the study period.
10. Any condition that may preclude the participant from completion of study related activities; such as planned travel, or out of the state of residence and not able to return for follow-up visits or relocation of residence.
11. Females of reproductive age unless proven to be urine HCG negative at the time of participation.
12. Recent opportunistic infection, such as CMV, EBV, BK viral reactivation, or any other documented or laboratory confirmed opportunistic infection or on treatment for confirmed infection.
13. Vulnerable subjects such as aged less than 18 years, pregnant women, nursing home residents or other institutionalized persons, students, employees, prisoners, and persons who may not be able to make independent decisions or is considered to have a cognitive impairment, or non-English speaking in the absence of a reliable interpreter or translator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravinder Wali, MD, Principal Investigator — Inova Fairfax Hospital
Locations (1):
- Inova Fairfax Hospital, Falls Church, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SD-IIV3: Standard-dose trivalent (SD-IIV3) flu vaccine
- HD-IIV3: high dose trivalent flu vaccine recipients
Period: Overall Study
Arm/Group | SD-IIV3 | HD-IIV3
Started | 30 | 32
Completed | 26 | 30
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- SD-IIV3: Standard-dose trivalent (SD-IIV3) seasonal influenza vaccine
- HD-IIV3: high-dose trivalent (HD-IIV3) seasonal influenza vaccine
- Total: Total of all reporting groups
Arm/Group | SD-IIV3 | HD-IIV3 | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 26 | 53
  >=65 years | 3 | 6 | 9
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 54.9 [45.75 to 64.25] | 56.6 [53 to 63.25] | 55.7 [49.5 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 20
  Male | 23 | 19 | 42
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Local Site Reactions
Description: Evaluation of local and systemic reactions, use of analgesics or antipyretics.
Time Frame: Day 1 and weeks 1, 4, and 12
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Flu Vaccine | Flu Vaccine
Number analyzed (Participants) | 32 | 30
Participants | 2 | 2

2. Primary Outcome: Measurement of Strain-specific Hemagglutination Inhibition (HI) Antibody Titers
Description: Number of patients and percentage of subjects achieving hemagglutination inhibition (HI) titer≥40
Time Frame: Week 1, 4, and 12
Measure: Count of Participants; unit: Participants
Groups:
- SD-IIV3: Standard dose flu vaccine
- HD-IIV3: high dose flu vaccine
Arm/Group | SD-IIV3 | HD-IIV3
Number analyzed (Participants) | 30 | 32
Participants
  week 1 | 14 | 19
  Week 4 | 16 | 23
  Week 12 | 15 | 21

3. Secondary Outcome: All Cause ED Visits/Unscheduled Clinic Visits
Description: All-cause outpatient/Emergency department visits during study follow-up (other than pre-specified post transplant follow-up visits).
Time Frame: day 1 - 3 months
Measure: Count of Participants; unit: Participants
Groups:
- High Dose Flu Vaccine (HD-IIV3): influenza trivalent inactive vaccine high dose. IM (intramuscular) injection one time administration
  influenza trivalent inactive vaccine high dose: one time IM injection of high dose influenza vaccine to measure immunogenicity, safety, and efficacy in organ transplant recipients
- Standard Dose (SD-IIV3): influenza trivalent inactive vaccine IM injection one time administration
  influenza trivalent inactive vaccine: one time IM injection of standard influenza vaccine to measure immunogenicity, safety, and efficacy in organ transplant recipients
Arm/Group | High Dose Flu Vaccine (HD-IIV3) | Standard Dose (SD-IIV3)
Number analyzed (Participants) | 32 | 30
Participants | 30 | 25

4. Secondary Outcome: Number and Percentage of Subjects in Each Group Achieving Seroconversion for Each Strain
Description: Number and percentage of subjects in each group achieving seroconversion (at least 4-fold increase in titers from baseline) for each any strain at weeks 4 and 12
Time Frame: Week 4 and Week 12
Population: Analysis performed only for participants between ages of 18 and 65.
Measure: Count of Participants; unit: Participants
Groups:
- Standard Dose Flu Vaccine: standard influenza trivalent inactive vaccine dose. IM (intramuscular) injection one time administration
- High Dose Flu Vaccine: influenza trivalent inactive vaccine IM injection one time administration
Arm/Group | Standard Dose Flu Vaccine | High Dose Flu Vaccine
Number analyzed (Participants) | 27 | 26
Participants
  week 4 | 7 | 6
  week 12 | 7 | 7

ADVERSE EVENTS:
Groups:
- SD-IIV3: The safety and immunogenicity of seasonal influenza vaccination using Standard-dose trivalent (SD-IIV3) in recipients of solid organ transplants who were at least 30 days after transplantation via a randomized blinded study.
- HD-IIV3: The safety and immunogenicity of seasonal influenza vaccination using high-dose trivalent (HD-IIV3) in recipients of solid organ transplants who were at least 30 days after transplantation via a randomized blinded study.
Arm/Group | SD-IIV3 | HD-IIV3
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 13/30 | 14/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SD-IIV3 (N=30) | HD-IIV3 (N=32)
local pain (Musculoskeletal and connective tissue disorders) | 13 | 13
redness (General disorders) | 8 | 12
swelling (General disorders) | 13 | 14
fever (General disorders) | 10 | 10
headache (General disorders) | 9 | 9
fatigue (General disorders) | 7 | 11
nausea, vomiting, diarrhea (General disorders) | 5 | 9
myalgia (General disorders) | 10 | 9
arthralgia (General disorders) | 10 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No